CLINICAL TRIAL: NCT00508963
Title: Compassionate Use of Sodium Stibogluconate (Pentostam) for Cutaneous and Mucocutaneous New World Leishmaniasis
Status: No longer available | Type: Expanded Access
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF Infectious Diseases
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-05

CONDITIONS: Leishmaniasis, Cutaneous; Leishmaniasis, Mucocutaneous
Keywords: New World Cutaneous or Mucocutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis, Mucocutaneous | interventions — Antimony Sodium Gluconate

INTERVENTIONS:
Drug: sodium stibogluconate (Pentostam) — 20 mg/kg IV every day for 20 or 28 days

SUMMARY:
Patients with biopsy proven new world cutaneous or mucocutaneous leishmaniasis will be treated with sodium stibogluconate (Pentostam).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven new world cutaneous or mucocutaneous leishmania

Exclusion Criteria:

* Prolonged QT
* Liver disease
* Pancreatitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schwartz, MD, Principal Investigator — University of CA at San Francisco; Kanade Shinkai, MD, Principal Investigator — University of CA at San Francisco
Locations (1):
- University of CA at San Francisco Hospitals and Clinics, San Francisco, California, United States